CLINICAL TRIAL: NCT05024448
Title: Glucocorticosteroid Treatment in Acute Unilateral Vestibulopathy, a Multicentric, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Glucocorticosteroid Treatment in Acute Unilateral Vestibulopathy (Vestibular Neuronitis)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Nils Guinand, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB_2020-00001
Record Dates: First submitted 2021-07-28; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Acute Peripheral Vestibulopathy
MeSH Terms: conditions — Vestibular Neuronitis | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone (Active Comparator): Prednisone, 60mg/d, for 10 days
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — oral administration, 60mg/d for 10d

SUMMARY:
The vestibular system is a part of the inner ear and functions as a motion sensor. It provides the central nervous system with information about changes of the head position. This information is essential for the proper functioning of the balance system. In particular, it ensures effective postural control and gaze stabilization. Abrupt vestibular deficit is defined as a sudden loss of the vestibular function. In the acute phase the patient presents mainly with intense rotatory vertigo and instability, most often accompanied by nausea. The symptoms are exacerbated by head movements. The diagnosis is made by observation of a spontaneous nystagmus, measurement of a pathological head impulse test and an asymmetric response to caloric tests, in the absence of other neurological symptoms. Although the etiology is unknown, it could be of viral or vascular origin. Symptoms usually regress within a few days or weeks. Vestibular function recovers in about half of the cases, in the other half a central compensation process is set up. The benefit of a 3-week course of corticosteroids has been demonstrated in one study. The dosage has been debated. The aim of this study is to demonstrate the benefit of a 10-day course of oral corticosteroids. The primary objective is to demonstrate a significant reduction in the rate of asymmetry of caloric response and the secondary objective is to demonstrate a significant reduction in the impact of symptoms assessed with the Dizziness Handicap Inventory (DHI) score at 1 year.

ELIGIBILITY:
Inclusion Criteria:

Medical History :

* severe and prolonged rotatory vertigo;
* acute onset, subacute, within 3 days;
* nausea ;
* imbalance.

Physical examination :

* spontaneous nystagmus beating towards the healthy ear (fast phase);
* no evidence of central vestibular lesion;
* Head impulse test abnormal, at least for the lateral semicircular canal (in some cases, the sign is only detectable for the 2 vertical semicircular canals with specific equipment, mostly not available in current practice);
* areflexia or hyporeflexia (asymetry > 70% calculated according to the classical Jongkees formula [slow phase velocity of the nystagmus in response to caloric stimulation at (right at 30°C + right at 44°C) - ( left at 30°C + left at 44°C ) / (right 30°C + left 30°C + right 44°C + left at 44°C) x 100], in the caloric test (10 cc in 20 s, at 30 and 44° C)

Exclusion Criteria:

* history of vestibular disorders other than benign paroxysmal positionning vertigo (BPPV);
* symptoms lasting more than 3 days;
* cochlear symptoms (deafness before, during or after vertigo);
* central oculomotor dysfunction;
* central vestibular dysfunction;
* signs of brain dysfunction (e.g. epilepsy);
* MRI (if done) abnormal central vestibular pathways;
* psychiatric disease (history of psychiatric disease);
* glaucoma ;
* acute infection (herpes simplex, herpes zoster, corneal herpes, chicken pox, tuberculosis);
* patients already on corticosteroids;
* severe diabetes (fasting blood glucose > 7 mmol/l);
* Severe hypertension (systolic >180; diastolic > 110);
* contraindications to glucocorticoids (peptic ulceration, osteoporosis confirmed by bone density tests or pathological fractures);
* allergy to glucocorticoids or mannitol
* malignant disease;
* cardiac disease (recent myocardial infarction, heart failure);
* liver dysfunction (cirrhosis)
* renal insufficiency;
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Bithermal calorics asymetry | Day 1
Bithermal calorics asymetry | Day 21
Bithermal calorics asymetry | Day 365

SECONDARY OUTCOMES:
Dizziness Hanidcap Inventory (Questionnaire) | Day 1, Day 21, Day 365
  min: 0 / max:100, higher score is worse

IPD SHARING:
Plan to Share IPD: No